CLINICAL TRIAL: NCT00517296
Title: EUS Guided Treatment With Humira for Crohn's Perianal Fistulas
Brief Title: Endoscopic Ultrasound (EUS) Guided Treatment With Humira for Crohn's Perianal Fistulas
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, David Schwartz, Principal Investigator, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 061178
Record Dates: First submitted 2007-08-15; First posted 2007-08-16 (Estimated); Results first posted 2017-04-21 (Actual); Last update posted 2017-04-21 (Actual); Status verified 2017-03

CONDITIONS: Crohn Disease; Rectal Fistula
MeSH Terms: conditions — Crohn Disease; Rectal Fistula | interventions — Emergency Use Authorization; Adalimumab

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Surgeon did not have access to EUS data for the control group prior to exam under anesthesia (EUA) and surgical intervention.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adalimumab with EUS guided therapy (Experimental): Patients will be randomized to adalimumab treatment with EUS guided therapy decisions. Colorectal surgeon will have access to EUS data prior to EUA with possible seton placement.
  Interventions: Procedure: EUA with seton placement if necessary; Drug: adalimumab; Procedure: EUS
- Adalimumab (Active Comparator): Patients will be randomized to adalimumab treatment. Colorectal surgeon will not have access to EUS data prior to EUA with possible seton placement.
  Interventions: Procedure: EUA with seton placement if necessary; Drug: adalimumab

INTERVENTIONS:
Procedure: EUA with seton placement if necessary — Patients randomized to the combination therapy group, the surgeon will have access to EUS findings.
Drug: adalimumab — Patients began therapy with adalimumab using clinic standards for dosing.
Procedure: EUS — Patients in combination therapy group had an EUS done every 12 weeks to help guide therapy.
  Arms: Adalimumab with EUS guided therapy

SUMMARY:
This study is to assess whether utilizing endoscopic ultrasound(EUS) to guide treatment can improve durable fistula healing in patients with Crohn's perianal fistulas and to get preliminary information regarding the effectiveness of Adalimumab for Crohn's perianal fistulas.

DETAILED DESCRIPTION:
Prospective randomized trial to assess the effectiveness of rectal EUS to guide perianal fistula treatment. Our hypothesis is that using imaging, in this case endoscopic ultrasound (EUS), to initially evaluate and then guide therapy with an anti-TNF agent (adalimumab) for fistulizing disease will lead to better short- and long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

A patient may be considered for study participation if all of the following apply:

* Male and Female aged 18 years or older; and
* A confirmed diagnosis of Crohn's disease and one or more identifiable perianal fistulas.

Exclusion Criteria:

A patient will be excluded from the study if one or more of the following apply:

* Females who are pregnant or breast feeding;
* Infliximab received within 6 weeks prior to study entry;
* Patients who cannot take, or refuse to take concomitant immunosuppressive therapy with either azathioprine, 6-mercaptopurine, or methotrexate; Unless patient has been intolerant of these therapies in the past or is contraindicated as determined by the investigator;
* Patients who cannot take, or refuse to take concomitant antibiotic therapy;
* Patients with severe anal stenosis or tenderness which would preclude colonoscopy and / or rectal EUS;
* Patients who cannot take or refuse to take adalimumab;
* Patients with active or latent tuberculosis;
* Patients who have had systemic antibiotic, antiviral or antifungal treatment(s) within 3 weeks prior to Screening for all non-Crohn's related infections;
* Patients concurrently taking anakinra (Kineret);
* Patients with a history of cancer or lymphoproliferative disease other than a successfully and completely treated cutaneous squamous cell or basal cell carcinoma or carcinoma in-situ of the cervix;
* Patients with chronic hematologic problems such as bleeding dyscrasias;
* Patients with a history of demyelinating disease (i.e. multiple sclerosis); and
* Patients with congestive heart failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-01; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A Schwartz, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Adalimumab With EUS Guided Therapy | Adalimumab
Started | 10 | 11
Completed | 9 | 11
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adalimumab With EUS Guided Therapy | Adalimumab | Total
Number analyzed (Participants) | 9 | 11 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 11 | 20
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 9 | 11 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Durable Fistula Healing
Description: Complete cessation of fistula drainage at 48 weeks
Time Frame: at week 48
Measure: Number; unit: participants
Arm/Group | Adalimumab With EUS Guided Therapy | Adalimumab
Number analyzed (Participants) | 9 | 11
participants | 7 | 8

2. Secondary Outcome: Changes in Disease Activity
Description: Changes in Crohn's disease activity using the Harvey Bradshaw Index (HBI) at Week 48 compared to baseline HBI Scores. Higher numbers for the HBI equal more significant disease activity. Range can vary from 0 to 17 plus the number of liquid stools per day.
Time Frame: Baseline and 48 Weeks
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Arm/Group | Adalimumab With EUS Guided Therapy | Adalimumab
Number analyzed (Participants) | 9 | 11
units on a scale | -5.0 [-7.5 to -3.0] | -1.0 [-9.0 to 0.0]

3. Secondary Outcome: Changes in Perianal Disease Activity Index (PDAI)
Description: Changes in Crohn's disease activity at Week 48 compared to baseline based on PDAI Scores- higher numbers equal more significant disease activity. PDAI has a range from 0 to 20.
Time Frame: Baseline and 48 Weeks
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Arm/Group | Adalimumab With EUS Guided Therapy | Adalimumab
Number analyzed (Participants) | 9 | 11
units on a scale | -5.50 [-6.00 to -5.00] | -5.0 [-7.25 to -3.5]

ADVERSE EVENTS:
Time Frame: Adverse events were captured beginning with date of consent and continuing through final study visit (week 48). If an adverse event was ongoing at the time of study completion, the event was followed until resolved.
Groups:
- A, Combination Therapy Group: Group A patients will be randomized to TNF and seton placement.
  Seton placement: Patients randomized to the combination therapy group will have seton placement prior to initiating therapy with Certolizumab.
- B, Control Arm: Group B patients will be randomized to surgical guidance / standard of care
Arm/Group | A, Combination Therapy Group | B, Control Arm
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/11
Other Adverse Events (participants affected / at risk) | 3/9 | 1/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A, Combination Therapy Group (N=9) | B, Control Arm (N=11)
Incision and draining procedures of abscess (Gastrointestinal disorders) | 3 (3) | 1 (1) — Incision and drainage procedure and placement of setons for a new abscesses that developed during treatment based on clinical assessment (control group) or imaging (eus group)

LIMITATIONS AND CAVEATS:
Small sample size which increases the chance of type II error.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes